CLINICAL TRIAL: NCT07131826
Title: The Quality of Life and Viral Control Effect of AIDS Patients After Long-acting Injection of Cabotegravir and Rilpivirine
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Clinical Trial Center (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor-Investigator, National Taiwan University Clinical Trial Center, WANG-HUEI SHENG professor, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Other Study IDs: 202503037RINA
Record Dates: First submitted 2025-04-28; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-04

CONDITIONS: Viral Control; Quality of Life; Cabotegravir; Rilpivirine; AIDS
Keywords: cabotegravir; rilpivirine; AIDS; quality of life; viral control
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AIDS patients after long-acting injection of cabotegravir and rilpivirine: AIDS patients after long-acting injection of cabotegravir and rilpivirine
  Interventions: Other: Observational study, non-interventional

INTERVENTIONS:
Other: Observational study, non-interventional — Observational study, non-interventional

SUMMARY:
"AIDS" was once regarded as the Black Death of the 20th century. However, with the advent of cocktail therapy, the survival rate of infected people has been greatly improved and the average life expectancy has been increased. Today, AIDS is considered a chronic disease, just like hypertension and diabetes. As long as you have regular checkups and take medication on time every day, you can complete the treatment, just like a normal person. However, there is still a risk of missing medication when taking it every day, and long-term missed medications can easily lead to drug resistance and increase the risk of treatment failure. After the HIV-infected person has stabilized the viral load, their mobility, self-care and daily activities are no different from those of normal people. However, they experience side effects such as fatigue, lack of energy, difficulty sleeping, depression, changes in appearance, tension and anxiety, dizziness, headache, vomiting, etc., which affect their quality of life. The long-acting AIDS injection is a long-acting dosage form for intramuscular injection. It has been included in the national health insurance reimbursement standards. Treatment with long-acting injections can reduce the risk of infected people forgetting to take medicine, and there is no need to worry about the exposure of the disease when storing the medicine. Through this study, we hope to collect the results of long-acting injections for stable HIV treatment cases (health status, daily activities, injection site, satisfaction), and confirm that long-acting injections can significantly improve the quality of daily life of HIV-infected people.

ELIGIBILITY:
Inclusion Criteria:

18 years and above Clinical diagnosis of HIV infection completed long-acting injectable treatment Accept the questionnaire

Exclusion Criteria:

Not clinical diagnosis of HIV infection Do not accept questionnaires

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females aged 18 years or older who have completed long-acting injectable treatment for HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To whether long-acting injections can significantly improve the quality of daily life of people infected with HIV using a questionnaire | From the date of approval by the CTC to December 31, 2026.

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Does the long-acting injection improve the quality of daily life of HIV-infected people?
Supporting Information: Study Protocol